CLINICAL TRIAL: NCT00003076
Title: Phase IIb Chemoprevention Trial of Difluoromethylornithine (DFMO) in Human Subjects With Intestinal-type Barrett's Esophagus
Brief Title: Eflornithine to Prevent Cancer in Patients With Barrett's Esophagus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Prevention
Other Study IDs: CDR0000065763; P30CA046592 (NIH); CCUM-9555 (Other: University of Michigan Cancer Center PRC); NCI-P97-0094
Record Dates: First submitted 1999-11-01; First posted 2004-04-23 (Estimated); Last update posted 2012-12-19 (Estimated); Status verified 2012-12

CONDITIONS: Esophageal Cancer
Keywords: esophageal cancer
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Eflornithine

INTERVENTIONS:
Drug: eflornithine

SUMMARY:
RATIONALE: Chemoprevention therapy is the use of drugs to try and prevent the development or recurrence of cancer. It is not known whether eflornithine is effective in preventing cancer in patients with Barrett's esophagus.

PURPOSE: Randomized double-blinded phase II trial to study the effectiveness of eflornithine in preventing cancer in patients with Barrett's esophagus.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine whether oral eflornithine (DFMO) given in this study will cause significant reduction of the Ki67 labelling index in subjects with intestinal type Barrett's esophagus and low grade dysplastic Barrett's esophagus. II. Determine whether oral DFMO will alter the pathology and morphology of Barrett's esophagus. III. Determine whether there is a difference in cellular DNA ploidy and/or nuclear or nucleolar morphometry in patients with dysplastic Barrett's esophagus and nondysplastic intestinal type Barrett's esophagus compared to normal gastric fundic mucosa. Determine whether DFMO modulates changes in these surrogate endpoint biomarkers towards normal mucosal values. IV. Determine whether cells demonstrating nuclear p53 protein accumulation are either lost or undergo a change in cellular distribution, following treatment of patients with dysplastic Barrett's mucosa with DFMO. V. Determine whether DFMO modulates changes in growth factor or oncogene expression in dysplastic Barrett's esophagus and nondysplastic intestinal type Barrett's esophagus. VI. Determine whether pathologic or biologic surrogate modulation occurring during 6 months of DFMO treatment reverts 6 months after treatment is discontinued.

OUTLINE: This is a randomized, placebo controlled, double blind prevention study. Patients are initially stratified by dysplasia status at baseline (metaplastic vs low grade dysplastic) and treatment group (placebo vs eflornithine). Patients are randomized to receive daily doses of eflornithine (DFMO) or placebo for 26 weeks. At 0, 4, 8, 12, 16, 20, and 26 weeks there are toxicity and adherence evaluations and at weeks 26 and 52 patients have follow-up endoscopies.

PROJECTED ACCRUAL: A total of a 152 evaluable patients will be accrued in this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Must have a columnar lined esophagus that meets the following criteria: Specialized intestinal metaplasia Nondysplastic or low grade dysplasia Extends a minimum of 1 cm above the gastroesophageal junction

PATIENT CHARACTERISTICS: Age: Over 18 Performance status: Karnofsky 80-100% Life expectancy: Not specified Hematopoietic: WBC greater than 4,000/mm3 Platelet count greater than 120,000/mm3 Hemoglobin greater than 12 g/dL Prothrombin time less than 3 seconds beyond control Partial thromboplastin time less than 10 seconds beyond control Hepatic: Bilirubin less than 1.5 mg/dL Transaminases less than 1.5 times normal Renal: Creatinine less than 1.5 mg/dL Urinalysis: less than 1+ protein, 0-3 urinary casts, 0-5 white blood cells and red blood cells Cardiovascular: No severe dyspnea at rest, orthopnea, edema, history of congestive heart failure requiring continued treatment, or unstable angina Neurologic: No severe degenerative neurologic disease Pulmonary: No requirement of supplemental oxygen for exertion or rest Other: No prior malignancy within 5 years No active rheumatoid arthritis, lupus or other rheumatologic autoimmune disease (no less than 2 years of quiescence if inactive) No history of abnormal wound healing No history of esophageal varices or variceal bleeding Not pregnant or nursing Negative pregnancy test Adequate contraception required of all fertile patients

PRIOR CONCURRENT THERAPY: No regular, scheduled use of antiinflammatory medications, steroids, or anticoagulants No nutritional supplements other than two multivitamins per day or four single nutrient vitamin supplements per day

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Estimated)
Dates: Start 1995-10; Primary Completion 2002-06 (Actual); Study Completion 2005-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dean E. Brenner, MD, Study Chair — University of Michigan Rogel Cancer Center
Locations (5):
- United States (5):
  - Tulane University School of Medicine, New Orleans, Louisiana
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Arthur G. James Cancer Hospital - Ohio State University, Columbus, Ohio
  - Veterans Affairs Medical Center - Dallas, Dallas, Texas